CLINICAL TRIAL: NCT02798562
Title: Evaluation of the High-resolution, Contrast Enhanced Low-dose Breast-CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-135
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: BI-RADS 4; BI-RADS 5; BI-RADS 6; High Risk of Breast Cancer Which Indicates a Mamma-MRI
Keywords: low dose CT; contrast-enhanced; breast cancer screening; computer tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Native and dynamic contrast-enhanced CT (Experimental): Patients will undergo a native high-resolution and a dynamic contrast-enhanced CT, both sides respectively.
  Interventions: Device: Native and dynamic contrast-enhanced CT

INTERVENTIONS:
Device: Native and dynamic contrast-enhanced CT

SUMMARY:
The aim of this study is the clinical establishment of a native and contrast-enhanced computer tomography of the breast. The early detection of breast cancer is still a great challenge. Even though the implementation of the digital mammography combined with the mandatory screening-programs lead to significant improvements, sensitivity and specificity of these examinations need to be clearly classified as improvable. Generally, it is stated that the necessary transit from 2-D projected images to 3-D tomography will be crucially advantageous as magnetic resonance imaging has already shown. Similar or even major advantages can be expected by new approaches regarding CT with very high local resolution, better than 100µm in 3D and lower dose, under 5 Milligray (mGy), as demanded for a screening. A device that meets these demands and is also applicable for dynamic scans after intravenous administration of a contrast agent, has been developed with the support by the European Union (EU), German Research Foundation (DFG) and Federal Ministry of Education and Research (BMBF). Publications on technical and experimental results are already available. An evaluation in the clinical use is missing yet. The primary aim of this study is to evaluate systematically the performance of the native and dynamic, contrast-enhanced CT of the breast.

ELIGIBILITY:
Inclusion Criteria:

Sub Study 1:

* patients with mammographic or sonographic validated Breast Imaging Reporting and Data System (BI-RADS)-4 or BI-RADS-5-result or in BI-RADS-6-situation, i.e. with an already reliable carcinoma by punch biopsy, for which a clinical indication for a mamma-MRI consists.
* Age >= 40
* maintained renal function (MDRD with GFR >= 60 ml/min/1,73m²)
* normal thyroid function, no clinical indication for an endocrine autonomy, normal TSH (not older than 8 weeks)
* Persons which are able to give written consent and are aware of the nature, meaning and extent of the study
* signed informed consent

Substudy 2:

* patients with a doubtful and suspect clinical or mammographic or sonographic result (BI-RADS 3, 4a, 4b, 4c, 5) as well as patients with a reliable carcinoma by punch biopsy (BI-RADS 6), patients with high risk of breast cancer for which a clinical indication for a mamma-MRI consists.
* Age >= 40
* maintained renal function (MDRD with GFR >= 60 ml/min/1,73m²)
* normal thyroid function, no clinical indication for an endocrine autonomy, normal TSH (not older than 8 weeks)
* Persons which are able to give written consent and are aware of the nature, meaning and extent of the study
* signed informed consent

Exclusion Criteria:

Substudy 1:

* Pregnancy or lactation
* Women with child-bearing potential without sufficient contraception
* Age <40 years
* Women with proven pathogenic Breast Cancer (BRCA) 1-mutation or heterozygote risk (>= 25%)
* Hospitalization of patient ordered by the court or local authorities
* Relationship of dependence or employment to sponsor or investigator

additionally the following criteria apply, if conducting the dynamic contrast-enhanced breast-CT

* signs of a renal insufficiency (GFR < 60ml/min/1,73m²)
* clinical signs or signs of the labor chemistry for endocrine autonomy (increase of TSH)
* Patients with known allergies or intolerance reactions grade II or higher to contrast medium containing iodine

Substudy 2:

* Pregnancy or lactation
* Women with child-bearing potential without sufficient contraception
* Age <40 years
* Women with proven pathogenic BRCA 1-mutation or heterozygote risk (>= 25%)
* Hospitalization of patient ordered by the court or local authorities
* Relationship of dependence or employment to sponsor or investigator

additionally the following criteria apply, if conducting the dynamic contrast-enhanced breast-CT:

* end stage or advanced renal insufficiency
* clinical signs or signs of the labor chemistry for endocrine autonomy (increase of TSH)
* Patients with known allergies or intolerance reactions grade II or higher to contrast medium containing iodine

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Sub-Study 1: comparison of a-posteriori sensitivity using the native, contrast-enhanced or dynamic contrast-enhanced breast CT. | 2 years
  By using the images diagnostic criteria for identification and characterization of the pathologic and physiologic changes of the female breast will be elaborated.

SECONDARY OUTCOMES:
Comparison of biological value of the diagnosed carcinoma in dependence with its detection mode. | 2 years
  Detection mode means the prospective visibility of a carcinoma in one or more independent imaging methods, respectively.
  Biological value will be calculated by amount of high and intermediate grade vs. low grade lesions, status of Ki-67 values, distribution of luminal a, luminal b, Her2/neu and basal, distribution of receptor status
Substudy 2: sensitivity of the native and the contrast-enhanced or dynamic contrast-enhanced high-resolution low-dose CT in comparison to the conventional examination procedures | 2 years
Sub-study 2: specificity of the native and the contrast-enhanced or dynamic contrast-enhanced high-resolution low-dose CT in comparison to the conventional examination procedures | 2 years
Substudy 2: Positive Predictive Value (PPV) of the native and the contrast-enhanced or dynamic contrast-enhanced high-resolution low-dose CT in comparison to the conventional examination procedures | 2 years
Substudy 2: Negative Predictive Value (NPV) of the native and the contrast-enhanced or dynamic contrast-enhanced high-resolution low-dose CT in comparison to the conventional examination procedures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kuhl, Univ.-Prof. Dr. med., Principal Investigator — Klinik für Diagnostische und Interventionelle Radiologie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigel M, Vollmar SV, Kalender WA. Spectral optimization for dedicated breast CT. Med Phys. 2011 Jan;38(1):114-24. doi: 10.1118/1.3523599. PMID 21361181
- [Background] Nowak T, Hupfer M, Althoff F, Brauweiler R, Eisa F, Steiding C, Kalender WA. Time-delayed summation as a means of improving resolution on fast rotating computed tomography systems. Med Phys. 2012 Apr;39(4):2249-60. doi: 10.1118/1.3697533. PMID 22482646
- [Background] Beister M, Kolditz D, Kalender WA. Iterative reconstruction methods in X-ray CT. Phys Med. 2012 Apr;28(2):94-108. doi: 10.1016/j.ejmp.2012.01.003. Epub 2012 Feb 10. PMID 22316498
- [Background] Kuhl C, Weigel S, Schrading S, Arand B, Bieling H, Konig R, Tombach B, Leutner C, Rieber-Brambs A, Nordhoff D, Heindel W, Reiser M, Schild HH. Prospective multicenter cohort study to refine management recommendations for women at elevated familial risk of breast cancer: the EVA trial. J Clin Oncol. 2010 Mar 20;28(9):1450-7. doi: 10.1200/JCO.2009.23.0839. Epub 2010 Feb 22. PMID 20177029
- [Background] Kuhl CK. The "coming of age" of nonmammographic screening for breast cancer. JAMA. 2008 May 14;299(18):2203-5. doi: 10.1001/jama.299.18.2203. No abstract available. PMID 18477789
- [Background] Kuhl CK, Schrading S, Bieling HB, Wardelmann E, Leutner CC, Koenig R, Kuhn W, Schild HH. MRI for diagnosis of pure ductal carcinoma in situ: a prospective observational study. Lancet. 2007 Aug 11;370(9586):485-92. doi: 10.1016/S0140-6736(07)61232-X. PMID 17693177